CLINICAL TRIAL: NCT05715502
Title: Assessment of the Toxicity of Focal Salvage Brachytherapy of Recurrent Prostate Cancer After Prior Radiotherapy - the Prospective Focal Salvage Brachytherapy Study (FocaSaBra)
Brief Title: Focal Salvage Brachytherapy Study (FocaSaBra)
Acronym: FocaSaBra
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FocaSaBra
Record Dates: First submitted 2022-12-13; First posted 2023-02-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: recurrence; prostate cancer; brachytherapy; focal treatment; salvage treatment; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Experimental: All recruited participants will be treated with salvage partial (focal) prostate brachytherapy for the lesion of recurrent prostate cancer with appropriate margin.
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — Radiation: focal low dose rate or high dose rate brachytherapy for the lesion with appropriate margin, defined in magnetic resonance or positron emission tomography All recruited participants will be treated with interstitial brachytherapy for local recurrence of prostate cancer. The low dose rate of brachytherapy is used with a total dose of 145 Gy in the clinical target volume for participants after hypofractionated radiotherapy, a high dose rate brachytherapy as monotherapy or boost with external beam radiotherapy The high dose rate brachytherapy with two fractions of 13 Gy in the clinical target volume with a 3 to 14 days break is used after primary low dose rate brachytherapy or external beam radiotherapy alone.

SUMMARY:
The aim of this prospective phase II study is to evaluate the toxicity of salvage partial (focal) prostate brachytherapy in patients after prior radiotherapy (standard teleradiotherapy with / without brachytherapy, hypofractionated, self-reactive HDR / LDR brachytherapy) with local recurrence on the part of the prostate gland.

DETAILED DESCRIPTION:
Prostate cancer is the second most common cancer among men in Poland. Currently, a large number of diagnosed patients undergo radical radiotherapy. Despite the high effectiveness of treatment, some patients experience failures in the form of regional and / or distant metastases, most often in the form of isolated local recurrence. In patients with suspected local recurrence, we can decide on emergency treatment after PET, pelvic MRI with an assessment of the prostate gland, and after excluding metastases. The oncological(NCCN ) and urological (EUA) recommendations allow salvage surgical treatment, observation, palliative pharmacological castration, or treatment using salvage brachytherapy.

Salvage surgical treatment is associated with a 30-65% chance of cure in the top cancer centers in the world, and the risk of significant toxicity ranges from 17 to 48%.

Treatment with brachytherapy, due to the intra-tissue nature and the short therapeutic range of radiation, can deliver a high dose to the treated area despite prior radiotherapy treatment and exhaustion of tolerance doses in critical organs, e.g., rectum and/or bladder. Treatment of the entire prostate gland gives a chance of disease-free survival for five years in approximately 65% of patients, according to the prospective study RTOG 0526. However, emergency treatment in this study was associated with a 14% risk of significant post-treatment toxicity requiring medical intervention. There are some reports in the literature on brachytherapy involving cancer in the part of the prostate gland (focal brachytherapy), but they are only retrospective. They show significant treatment efficacy and lower toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed by biopsy (fusion mapping biopsy preferred) recurrence of prostate cancer after prior radical radiotherapy (brachytherapy, external beam radiotherapy alone or with brachytherapy boost, stereotaxic radiotherapy)
* Localized tumor lesion assessed by MRI or in the case of MR contraindications with TRUS and CT
* Exclusion of distant metastases using CT, MR, or PET imaging
* PSA doubling time over six months
* PSA value <10 ng / ml
* No anti-androgen treatment in the year prior
* Dysuria on the IPSS (International Prostate Symptom Score) ≤ 20 points
* General condition according to the WHO scale ≤ 2
* Signing informed consent to participate in the study

Exclusion Criteria:

* PSA value> 10ng / ml
* General condition according to the WHO scale> 2
* Dysuria on the IPSS scale> 20 points
* PSA doubling time <6 months
* Inability to discontinue anticoagulants.
* An active urinary tract infection.
* Contraindications to general anesthesia
* Active inflammatory bowel diseases.
* Second active cancer or treatment with completion less than 3 years earlier, except for low-stage skin cancer
* Estimated Survival <5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change in the urological toxicity in points with the International Prostate Symptoms Scale | change from baseline to 24 months of follow-up
  Assessment of the change in the urological toxicity in points with the International Prostate Symptoms Scale - IPSS within 0-35 points
Assessment of the change in the erectile function in points with the International Index of Erectile Function 5 (IIEF-5) (0-25 points) | change from baseline to 24 months of follow-up
  Assessment of the change in the erectile function in points with the International Index of Erectile Function 5 (IIEF-5): scale 0-25 points
Assessment of the change in the quality of life in points with EORTC C30 and PR25 protocols. (0-100 points) | change from baseline to 24 months of follow-up
  Assessment of the change in the quality of life in points with EORTC C30 and PR25 protocols, scale: 0-100 points

SECONDARY OUTCOMES:
Assessment of the adverse events in the percentage of grades with the CTCAE v4.0 | 24 months after treatment
  Assessment of the adverse events in the percentage of grades with the CTCAE v4.0 scale: 0-5 grades

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Burchardt, PhD, MD, Principal Investigator — Greater Poland Cancer Centre / Brachytherapy Department
Locations (1):
- Greater Poland Cancer Centre / Brachytherapy Department, Poznan, Greater Poland Voivodeship, Poland

REFERENCES:
- [Background] Schaeffer E, Srinivas S, Antonarakis ES, Armstrong AJ, Bekelman JE, Cheng H, D'Amico AV, Davis BJ, Desai N, Dorff T, Eastham JA, Farrington TA, Gao X, Horwitz EM, Ippolito JE, Kuettel MR, Lang JM, McKay R, McKenney J, Netto G, Penson DF, Pow-Sang JM, Reiter R, Richey S, Roach Iii M, Rosenfeld S, Shabsigh A, Spratt DE, Teply BA, Tward J, Shead DA, Freedman-Cass DA. NCCN Guidelines Insights: Prostate Cancer, Version 1.2021. J Natl Compr Canc Netw. 2021 Feb 2;19(2):134-143. doi: 10.6004/jnccn.2021.0008. PMID 33545689
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Nguyen PL, D'Amico AV, Lee AK, Suh WW. Patient selection, cancer control, and complications after salvage local therapy for postradiation prostate-specific antigen failure: a systematic review of the literature. Cancer. 2007 Oct 1;110(7):1417-28. doi: 10.1002/cncr.22941. PMID 17694553
- [Background] Crook, J. M., Rodgers, J., Pisansky, T. M., Trabulsi, E., Amin, M., Bice, W., Morton, G., Pervez, N., Vigneault, E., Catton, C. N., Michalski, J. M., Roach, M., Beyer, D. C., Rossi, P. J., Horwitz, E. M., Donavanik, V., Sandler, H. M., Siva, S., Bressel, M., … Ball, D. (2020). Salvage Low Dose Rate Prostate Brachytherapy: Clinical Outcomes of a Phase II Trial for Local Recurrence after External Beam Radiotherapy (NRG/RTOG -0526). International Journal of Radiation Oncology, Biology, Physics, 108(3), S3. https://doi.org/10.1016/J.IJROBP.2020.07.2071
- [Background] Crook JM, Zhang P, Pisansky TM, Trabulsi EJ, Amin MB, Bice W, Morton G, Pervez N, Vigneault E, Catton C, Michalski J, Roach M 3rd, Beyer D, Jani A, Horwitz E, Donavanik V, Sandler H. A Prospective Phase 2 Trial of Transperineal Ultrasound-Guided Brachytherapy for Locally Recurrent Prostate Cancer After External Beam Radiation Therapy (NRG Oncology/RTOG-0526). Int J Radiat Oncol Biol Phys. 2019 Feb 1;103(2):335-343. doi: 10.1016/j.ijrobp.2018.09.039. Epub 2018 Oct 9. PMID 30312717
- [Background] Aaronson DS, Yamasaki I, Gottschalk A, Speight J, Hsu IC, Pickett B, Roach M 3rd, Shinohara K. Salvage permanent perineal radioactive-seed implantation for treating recurrence of localized prostate adenocarcinoma after external beam radiotherapy. BJU Int. 2009 Sep;104(5):600-4. doi: 10.1111/j.1464-410X.2009.08445.x. Epub 2009 Feb 23. PMID 19245439